CLINICAL TRIAL: NCT01145820
Title: Efficacy of Adjunctive Juice Plus in Reducing Post-operative Morbidity and Improving Quality of Life After Lower Third Molar Surgery: a Randomized Controlled Clinical Trial
Brief Title: Fruit And Vegetables and OUtcomes After Removal of Impacted TEeth
Acronym: FAVOURITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: NSA, Inc (Unknown)
Responsible Party: Principal Investigator, Thomas Dietrich, Dr. med., Dr. med. dent., MPH, Principle Investigator, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG_09-111
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Postoperative Morbidity; Trauma; Wound Healing
Keywords: third molar; trauma; pain; wound healing; post operative morbidity; acute trauma; short-term wound healing
MeSH Terms: conditions — Wounds and Injuries; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Juice Plus (Experimental)
  Interventions: Dietary Supplement: Juice plus
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Juice plus

INTERVENTIONS:
Dietary Supplement: Juice plus — Juice Plus (2 capsules bds) for 11 weeks (10 weeks preop and 1 week postop)

SUMMARY:
The proposed study will test the following hypotheses:

1. Pre-operative daily dual supplementation with Juice Plus+ (fruit & vegetable) for 11 weeks will result in reduced post-operative morbidity in terms of quality of life, pain and trismus after 1 week following surgical removal of lower third molars, when compared to placebo.
2. Pre-operative daily dual supplementation with Juice Plus+ (fruit & vegetable) for 11 weeks will reduce serum markers of oxidative stress, following surgical removal of lower third molars, when compared with placebo.

DETAILED DESCRIPTION:
In general antioxidant status appears to influence wound healing in humans and in animal models of acute trauma, with low antioxidant concentrations and excessive oxidative stress being associated with impaired healing. Whilst antioxidant supplementation has been reported to improve plasma antioxidant status and wound healing in animal models of acute trauma, there is remarkably little data from human studies.

The use of Juice Plus+ has been reported to increase serum concentrations of important antioxidants and reduce serum markers of oxidative stress. However, to date there are no reported studies concerning the potential for Juice Plus+ to improve patient-based outcome measures following the surgical removal of lower third molars. This study therefore proposes to investigate the impact of daily supplementation with Juice Plus+, in improving outcomes following surgical trauma. While the rationale for the proposed study is primarily predicated on the established role of oxidative stress and antioxidant micronutrients in chronic inflammatory diseases, the proposed randomized controlled clinical study represents an efficient way of evaluating the potential for adjunctive Juice Plus+ use in improving wound healing and reducing post-operative morbidity following surgical procedures on humans.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring surgical removal of a single (unilateral) mandibular wisdom tooth
2. Tooth requiring full mucoperiosteal flap to be raised for removal
3. Bone removal necessary during procedure.

Exclusion Criteria:

1. Patients refusing to give written informed consent
2. Clinically significant or unstable physical or mental disability rendering the participants incapable of complying with the study protocol as judged by the investigator
3. Pregnant or breast-feeding women
4. Patients taking long term anti-microbial or anti-inflammatory drugs
5. Patients unable to swallow Juice Plus capsules
6. Patients taking regular vitamin or mineral supplementation
7. Patients requiring pre-operative antibiotics for surgery
8. Patients requiring concomitant extractions or contralateral lower 3rd molar removal
9. Allergic to any of the ingredients contained in supplements or placebo medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 246 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life | first postoperative week
  QOL as assessed by PoSSe scale (Ruta et al., 2000)

SECONDARY OUTCOMES:
trismus | postoperative week
  trismus will be assessed by investigator at 48h and 1 week postoperative, and every postop day by patient
postoperative pain | postoperative week
  pain will be assessed by patient on VAS on each postop day. groups will be compared for the following:
  * total (sum) of pain scores over 1 week
  * proportion of patients reporting >50% pain on day 2 and day 7
  * time until pain consistently <50%
  * proportion of patients reporting 20mm increase in pain after postoperative day 3
analgesic use | first postoperative week
plasma total antioxidant capacity (TAOC) | baseline (preop) and 1 week postop
  group differences between plasma TAOC changes between baseline and 1 week postop
serum biomarkers of oxidative stress | first postoperative week (baseline and 1 week)
  differences in change from baseline to 1 week of mean protein carbonyls, isoprostanes and 8OHdG
serum concentration of acute phase reactants | first postoperative week
  change between baseline and 1 week of: CRP, fibrinogen, WBC
adverse events | first postoperative week

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietrich, DMD, MD, MPH, Principal Investigator — University of Birmingham; Iain Chapple, BDS, PhD, Principal Investigator — Unversity of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Gorecki P, Burke DL, Chapple ILC, Hemming K, Saund D, Pearson D, Stahl W, Lello R, Dietrich T. Perioperative supplementation with a fruit and vegetable juice powder concentrate and postsurgical morbidity: A double-blind, randomised, placebo-controlled clinical trial. Clin Nutr. 2018 Oct;37(5):1448-1455. doi: 10.1016/j.clnu.2017.08.004. Epub 2017 Aug 10. PMID 28866140